CLINICAL TRIAL: NCT00052325
Title: Iscar For Supplemental Care In Advanced Non-Small Cell Lung Carcinoma
Brief Title: Mistletoe in Treating Patients With Advanced Non-Small Cell Lung Cancer Who Are Receiving Palliative Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258166; TJUH-01F.45; TJUH-2001-35
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2005-07

CONDITIONS: Lung Cancer
Keywords: stage IV non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

INTERVENTIONS:
Dietary Supplement: mistletoe extract

SUMMARY:
RATIONALE: Mistletoe may help the body build an immune response and may improve quality of life to help patients live more comfortably.

PURPOSE: This phase II trial is studying mistletoe to see how well it works in treating patients who are receiving palliative chemotherapy for stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether supplemental treatment with mistletoe increases immune function (as determined by total lymphocyte count, eosinophil count, and lymphocyte subset analysis) in patients with stage IIIB or IV non-small cell lung cancer receiving palliative chemotherapy.
* Determine the tolerability of this drug in these patients.
* Correlate immune function and quality of life in patients treated with this drug.

OUTLINE: This is an open-label, non-randomized, multicenter study.

Patients receive mistletoe subcutaneously three times a week for 15 weeks.

Dose of mistletoe is increased at weeks 2 and 3 and then every 3 weeks until a maximum response is seen, dose-limiting toxicity occurs, or the study ends.

Quality of life is assessed at baseline and at weeks 3, 6, 9, 12, and 15.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Stage IIIB or IV non-small cell lung cancer

  * Newly diagnosed disease
* Planning to receive standard chemotherapy with either carboplatin plus paclitaxel or cisplatin plus gemcitabine

  * Refused or ineligible to participate in experimental chemotherapy clinical trials

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant
* No AIDS
* Able to self-report quality of life
* No known allergy to Viscum album Linnaeus

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent mistletoe products

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* No concurrent steroid or adrenocorticotropic hormone therapy

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent participation in other clinical trials
* No concurrent mushroom glucan or proteoglycan extracts
* No concurrent thymus extract
* No concurrent non-oncologic immunosuppressive therapy (e.g., therapy for rheumatoid arthritis or after organ transplantation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rosenzweig, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania, United States